CLINICAL TRIAL: NCT05094297
Title: Evaluating the Impact of Focused Muscle Contraction Therapy in U.S. Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Enrico Benedetti, Warren H. Cole Chair in Surgery, Professor and Head of Surgery, Medical Director, Abdominal Organ Transplant Program, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0832
Record Dates: First submitted 2021-09-20; First posted 2021-10-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Acute Pain; Fatigue; Depression
MeSH Terms: conditions — Chronic Pain; Acute Pain; Fatigue; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigate the effects of an exercise intervention on U.S. Veterans. (Experimental): A total of 25 U.S. Veterans (≥ 18 years of age), who suffer from pain, fatigue, low energy levels or are unable to physically do things they were once able to do, will be enrolled.
  Interventions: Behavioral: Investigate the effects of an exercise intervention on U.S. Veterans.

INTERVENTIONS:
Behavioral: Investigate the effects of an exercise intervention on U.S. Veterans. — Enrolled subjects will be asked to complete 94 total visits (4 study testing visits and 90 exercise visits). They will be tested for fitness, strength, and health risk factors at UIC 4 times and will complete 90 exercise training visits at the GH FITLab over the next 18 months.

SUMMARY:
This research study is being done to investigate if the GH Method exercise program positively affects body composition, improves physical abilities and can improve the overall sense of wellbeing (e.g. depression, PTSD, etc.) in U.S. Veterans. Subjects will be asked to complete 94 total visits (four (4) study testing visits and 90 exercise visits). Enrolled subjects will be tested for fitness, strength, and health risk factors at UIC 4 times and will complete 90 exercise training visits at the GH FITLab over the next 18 months. Subjects will also be asked to complete questionnaires about depression, post-traumatic stress symptoms and thoughts about harming oneself.

DETAILED DESCRIPTION:
The study will consist of 94 visits (4 study testing visits and 90 exercise visits). Subjects will come to UIC for study testing visits at baseline (prior to starting the exercise program), at 6 months, 12 months, and 18 months (after ending the exercise program). Each of those visits will take about 2-3 hours. After the initial baseline visit, subjects will come twice weekly, for roughly 1 hour each session, for 6 months (52 visits). From 6-12 months, subjects will come once a week, for roughly 1 hour each session (26 visits). From 12-18 months, subjects will come twice a month, for roughly 1 hour sessions (12 visits).

Methods:

Study Testing Visits

If subjects agree to be in the study, subjects will be asked to do the following procedures at baseline, 6 months, 12 months, and 18 months:

* Subjects will be asked to confirm their employment status each visit.
* Height and weight will be measured and body mass index (BMI) will be calculated.

Additionally, the investigators will measure the body fat composition and lean body mass using a DEXA scan.

* The investigators will ask subject's their age, race, number of injuries, number of fractures, surgical history, medical history, areas of pain, list of pain medications and allergies.
* Blood pressure will be measured for general health markers.
* Exercise limit will be measured with a timed 8 foot walk down the hallway (if applicable), a timed sit to stand test (sitting and standing 5 times in a row-if applicable), maximum sit to stands, and a balance test (standing in 3 different positions for 10 seconds each). These three tests combine to form a score called a short performance battery score.
* Strength and frailty will be measured using a grip dynamometer (squeezing a hand held device as hard as possible in their dominant hand three times.
* To evaluate general health, mental health (e.g. depression, post-traumatic stress disorder, etc.) and pain intensity, quality of life, measure of pain and disability, and fatigue, questionnaires will be administered.
* Subjects will be asked to disclose the number of hospital visits they have had in the last 18 months.
* Total weight lifted during training session will also be recorded.

Exercise Training Visits

After the initial baseline visit, subjects will begin their exercise training intervention which involves:

* Two days a week of exercise trainings for the first 6 months, and one day a week, from 6-12 months. From 12-18 months, subjects will then complete two days a month of exercise training. Each visit will last roughly one hour and will incorporate approximately 5-10 minute light warm-up plus stretching and then the exercises.
* At least twice weekly, GH Fitness staff will follow-up with subjects via text message, email or a phone call to evaluate subjects physical progress and overall health and energy.
* On Weeks 6, 13, 18, 25, 41, and 52 subjects will focus on cardio and endurance exercises. These exercises may include running in place, or using a recumbent (stationary) bike. All other weeks consist of basic strength training/resistance workouts.

List of All Possible Strength/Resistance Exercises

Exercise Chest: Smith Bench Press/Incline Glutes: Abductor Biceps: Cable Easy Curl/Free Bar Quads: Leg Extension Calves: Calf Machine Biceps: Preacher Quads: Leg Press Abs: Decline Back: Pull Down Behind Hamstring: Curl Machine Shoulders: Dumbbell Press / Smith Press Back: Low Roll Hamstring: Good Morning with Dumbbell/ 1 Leg Hamstring Curl Shoulders: Side Rise with Dumbbells Triceps: Push Down / Kick Back Abs: Sit Ups Triceps: Close Grip

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veterans
* Eligible subjects must be patients at the Jesse Brown VA Medical Center and suffer from pain, fatigue, low energy levels or are unable to physically do things they were once able to do.
* Subjects need to complete the PAR-Q with an acceptable score and/or must have written physician clearance.
* 18 years of age and older

Exclusion Criteria:

* Unable to travel to the training center
* Unable to give consent
* Unable to understand the study
* Unable to comply with the training program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate at which exercise will change body composition | 18 months
  With this hypothesis we will test whether muscle mass (DEXA scan) changes after 6 months, 12 months, 18 months of an exercise intervention. Baseline measurement will be performed before the intervention, at 6 months, 12 months, and at the end of the study (18 months) with muscle mass measured by DEXA.
Rate at which exercise will change body composition | 18 months
  With this hypothesis we will test whether muscle strength (dynamometer) changes after 6 months, 12 months, 18 months of an exercise intervention. Baseline measurement will be performed before the intervention, at 6 months, 12 months, and at the end of the study (18 months) with strength measured by dynamometer.

SECONDARY OUTCOMES:
Rate at which subjects will see changes in their physical abilities | 18 months
  We expect participants will see improvements in their physical abilities after 18 months in the exercise training sessions. This will be assessed by comparing baseline, 6 months, 12 months, and 18 months using a Short Physical Performance Battery test. This test requires the assessment of walking speed (time to walk 3 meters), a balance test (standing in 3 different positions for 10 seconds each-tandem, semi tandem, and side by side), and the time it takes to sit and stand 5 times in a chair (see above). Scoring is based on a scale of 0-12, lower numbers representing worse performance.
Rate at which subjects enrolled in the exercise intervention will have an overall changed sense of well-being. | 18 months
  Participants will be asked about their overall general health using the PROMIS.
Rate at which subjects enrolled in the exercise intervention will have an overall changed in fatigue. | 18 Months
  Participants will be asked about their mental health using the Fatigue Severity Index.
Rate at which subjects enrolled in the exercise intervention will have an overall changed in their quality of life. | 18 months
  Participants will be asked about their mental health using SF 36.
Rate at which subjects enrolled in the exercise intervention will have an overall decreased change in PTSD. | 18 months
  Participants will be asked about their mental health using the PSS-SR5.
Rate at which subjects enrolled in the exercise intervention will have an overall decreased change in depression. | 18 months
  Participants will be asked about their mental health using the BDI.
Rate at which subjects enrolled in the exercise intervention will have an overall change in pain intensity. | 18 months
  Participants will be asked about their overall pain intensity using the Numeric Rating Scale for Pain.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Benedetti, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No